CLINICAL TRIAL: NCT02800122
Title: PAthwAy of Dyspneic patIent in Emergency
Brief Title: PAthwAy of Dyspneic patIent in Emergency (PArADIsE)
Acronym: PArADIsE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHOUIHED Tahar (Other)
Collaborators: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor-Investigator, CHOUIHED Tahar, MD, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Other Study IDs: R2016-08
Record Dates: First submitted 2016-06-06; First posted 2016-06-15 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Dyspnea; Cardiac; Acute Disease
Keywords: acute dyspnea; emergency; acute heart failure
MeSH Terms: conditions — Dyspnea; Acute Disease; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with acute dyspnea: Patients with acute dyspnea treated by a medical team of emergencies of CHRU of Nancy.
  All patients admitted to the emergencies in the last 5 years matching the inclusion criteria will be evaluated. About 4,000 patients will be affected, including more than 800 patients with acute heart failure. (Figures based on export of ICD X codes (R06.0: Dyspnea) of patients cared in extra-hospital for acute dyspnea (diagnosis Dyspnea + Heart Failure) over the last 5 years).

SUMMARY:
This is an observational retrospective single-center study (CHRU of Nancy) in patients cared for acute dyspnea by a medical team of the emergencies of the CHRU of Nancy.

The main purpose of the study is to evaluate the outcome of patients cared for acute dyspnea by a medical team of emergencies of CHRU of Nancy.

DETAILED DESCRIPTION:
This observational retrospective single-center study will be conducted using data from medical records, acquired as part of usual care, patients cared for acute dyspnea in the last 5 years (from the date of authorization of data processing). About 4,000 patients will be affected, including more than 800 patients with acute heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Man or women ≥ 18 years
* Patients with acute dyspnea cared by a medical team of the emergencies of CHRU of Nancy.

Exclusion Criteria:

* Cardiorespiratory arrest before the care by a medical team of the emergencies of the CHRU of Nancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute dyspnea cared by a medical team of emergencies of CHRU Nancy in the last 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 24000 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
All cause in-hospital mortality | in the last 5 years

SECONDARY OUTCOMES:
Demographic and clinical data of patients cared by a medical team of emergencies | in the last 5 years
Duration of total hospitalization (including emergency stay and conventional hospitalization) | in the last 5 years
The main diagnosis of the initial hospitalization | in the last 5 years
Rate of Brain Natriuretic Peptide (BNP) | in the last 5 years
Administration of non-invasive ventilation and / or diuretics and / or nitrates | in the last 5 years
Administration time of non-invasive ventilation and / or diuretics and / or nitrates | in the last 5 years
Service type admitting the patient after the emergency care (intensive care, cardiology, intensive care cardiology, other ...) | in the last 5 years
Admission time in a service after the emergency care | in the last 5 years
Mortality and re-hospitalization of included patients | in the last 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tahar CHOUIHED, MD, PhD, Principal Investigator — Central Hospital, Nancy, France; Nicolas GIRERD, MD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- CHRU Nancy - Service des Urgences, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chouihed T, Bassand A, Duarte K, Jaeger D, Roth Y, Giacomin G, Delaruelle A, Duchanois C, Bannay A, Kobayashi M, Rossignol P, Girerd N. Head-to-head comparison of diagnostic scores for acute heart failure in the emergency department: results from the PARADISE cohort. Intern Emerg Med. 2022 Jun;17(4):1155-1163. doi: 10.1007/s11739-021-02879-6. Epub 2021 Nov 17. PMID 34787803
- [Derived] Chouihed T, Buessler A, Bassand A, Jaeger D, Virion JM, Nace L, Barbe F, Salignac S, Rossignol P, Zannad F, Girerd N. Hyponatraemia, hyperglycaemia and worsening renal function at first blood sample on emergency department admission as predictors of in-hospital death in patients with dyspnoea with suspected acute heart failure: retrospective observational analysis of the PARADISE cohort. BMJ Open. 2018 Mar 30;8(3):e019557. doi: 10.1136/bmjopen-2017-019557. PMID 29602842